CLINICAL TRIAL: NCT01009255
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of the H3 Receptor Antagonist, GSK239512 in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: Study to Evaluate the Efficacy and Safety of GSK239512 in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110651
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; placebo controlled; randomised; Histamine; H3 Antagonist; double blind; Cognition
MeSH Terms: conditions — Alzheimer Disease | interventions — GSK239512

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK239512 (Experimental): Oral tablets
  Interventions: Drug: GSK239512
- Placebo (Placebo Comparator): Placebo to match GSK239512.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK239512 — Histamine H3 Antagonist
  Arms: GSK239512
Drug: Placebo — Placebo to match GSK239512
  Arms: Placebo

SUMMARY:
This study aims to evaluate the cognitive enhancing effects and tolerability of GSK239512 compared to placebo in patients with mild to moderate Alzheimer's disease

DETAILED DESCRIPTION:
This is a 16-week, Phase II, multi-centre, randomised, double-blind, placebo-controlled, parallel group design study in male and female subjects with mild to moderate Alzheimers disease (AD). Subjects will undergo 2-week placebo run-in period before randomisation. They will undergo weekly review of safety, tolerability and cognitive performance measures.

ELIGIBILITY:
A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Male or female subjects with a clinical diagnosis of probable Alzheimer's disease in accordance with the NINCDS-ADRDA criteria, with symptoms of AD for at least 3 months.
* A Haschinski ischaemia score less than or equal to 4.
* Has undergone MRI or CT scan in the last 12 months. (For subjects not meeting this criteria, as scan will be conducted as part of the screening procedures).
* The subject has an MMSE score at Screening of 16 to 24 inclusive.
* Male or female aged 50 or above, at the time of signing the informed consent.
* If female, the subject must be post-menopausal, i.e. 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (<140 pmol/L) is confirmatory] or surgically sterile (documented tubal ligation or hysterectomy). [Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* The subject has the ability to comply with the study procedures as judged by the investigator.
* Subject lives with (or has substantial periods of contact with) a permanent caregiver who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status. A permanent caregiver is one who is able to provide care to the subject for the duration of the study without interruption for more than 1 week at a time. If at times during the study the permanent caregiver is unable to look after the subject, this period of absence of the caregiver must be covered by another caregiver. A permanent caregiver need not be living in the same residence with the subject. For such a caregiver, the investigator has to be satisfied that the subject can contact the caregiver readily during the times when the caregiver is not with the subject. If in doubt about whether a subject's care arrangements are suitable for inclusion, the investigator should discuss this with the GSK Medical Monitor.
* The subject has provided full written informed consent prior to the performance of any protocol specific procedure, or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative.
* The caregiver has provided his / her written consent prior to the performance of any protocol specific procedure
* AST and ALT less than 2xULN; alkaline phosphatase and bilirubin, less than or equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* If the subject is on any prior medications, they should satisfy the requirements in Section 9.

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* In the opinion of the investigator, following review of CT/MRI scans in the past 12 months and completion of neurological review there could be other probable causes of dementia which include, but are not limited to:
* History and/or evidence (CT or MRI scan performed since the onset of symptoms) of any other CNS disorder that could be interpreted as the primary cause of dementia: e.g. cerebrovascular disease, structural or developmental abnormality, epilepsy, infections, degenerative or inflammatory/demyelinating CNS conditions other than AD.
* Clinically significant focal findings on the neurological exam (excluding changes attributable to peripheral nervous system injury).
* Abnormal result of vitamin B12 and syphilis serology, where this is thought to be the cause of, or to contribute to the severity of, the subject's dementia. Subjects should be euthyroid based on laboratory results at the screening visit. Subjects maintained on thyroid medication must be euthyroid for a period of 2 months prior to the screening visit. If laboratory values are outside normal limits, but the investigator believes that the thyroid condition is stable and has no impact on cognition, such cases will be decided on case by case basis in discussion with the medical monitor.
* Diagnosis of possible, probable or definite vascular dementia in accordance with National Institute of Neurological Disorders and Stroke-Association Internationale pour la Recherche l'Enseignement en Neurosciences (NINDS-AIREN) criteria.
* Prior diagnosis of significant psychiatric illness such as schizophrenia or bipolar affective disorder with current symptoms related to the diagnoses such that in the opinion of the Investigator would interfere with participation in the study, or current depression (a score of greater than or equal to 8 on the Cornell Scale for Depression in Dementia), or subjects with other psychiatric features (including but not limited to having hallucinations) in their AD which in the opinion of the investigator, increase risk to safety.
* Subjects, who in the investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior in the last 6 months and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 2 months prior to screening.
* History or presence of significant sleep disturbance, such as severe insomnia or sleep disturbance associated with nocturnal wandering, nocturnal confusion / disorientation / agitation, which in the opinion of the investigator, may increase safety risk.
* History or presence of known or suspected seizures, unexplained significant loss of consciousness within last 6 months. Subjects who had febrile seizures in childhood may be included if these ceased by age 10 and they have had no other type of seizure in their medical history and have not been on anti-epileptic medications.
* History or presence of significant cardiovascular, gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, or any other clinically relevant abnormality, medical or psychiatric condition, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* History of alcohol or other substance abuse, according to the Diagnostic and Statistical Manual of Mental Disorders - Substance related disorders (DSM-IV) criteria within 3 years prior to the onset of AD symptoms, or since the onset of AD symptoms.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Uncontrolled hypertension with systolic BP greater than or equal to 160 and/or diastolic greater than or equal to 95 mmHg. Subjects with controlled hypertension with systolic BP less than 160 mmHg and diastolic less than 95 mmHg for at least 4 weeks are acceptable.
* Systolic BP less than 100 mmHg and/or diastolic less than 60 mmHg.
* Subjects with a QTcB and/or QTcF of greater than 450ms or greater than 480ms if they have bundle branch block or other ECG abnormalities which, in the opinion of the investigator is clinically significant in that they may increase safety risk.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Treatment with cholinesterase inhibitors (including Tacrine), memantine or selegiline within the last 3 months prior to screening. No patients with AD who are already on these medications at the time of screening will be recruited, as it would be unethical to withdraw these medications for study participation. Only AD subjects who are not yet on these medications, or who have withdrawn from these medications for other reasons previously, may be enrolled into this study.
* Use of the following medications within the last 30 days or 5 half-lives of these medications from screening (prohibited in Section 9.2):
* Any other treatments approved in the countries for treatment of cognitive symptoms of AD.
* Anti-psychotic drugs (typical or atypical dopaminergic antagonists or modulators).
* Any CNS stimulants (e.g., modafinil).
* Mood stabilization drugs (e.g. lithium, valproate, cabamazepine).
* Barbiturates, MAO inhibitors, Gingko biloba and other herbal treatments for cognitive impairment.
* Potent P-glycoprotein inhibitors (e.g. itraconazole, ketoconazole, cyclosporin, loperamide, diltiazem, verapamil, spironolactone, quinidine, bepridil, quinine, carvedilol).
* Known potent inhibitors or inducers of the CYP3A4 enzyme (e.g., verapamil, ketoconazole, cimetidine, rifampin, modafinil).
* Anti-cholinergic drugs or drugs which have anti-cholinergic effects (e.g. amitriptyline, amantidine).
* Anti-histamines which are CNS penetrant.
* Chronic sedative medications (greater than or equal to 4 days per week for the past 4 weeks prior to screening).
* Any other investigational drug.
* Use of other prescription or non-prescription drugs, including herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety, or are permitted under Section 9).
* Subjects who plan to commence treatment with prohibited medications in Section 9.2.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until the follow-up visit.
* Subjects who have commenced or are already undertaking a cognitive rehabilitation programme within 1 month of screening. Subjects who have stopped their cognitive rehabilitation programme at least 1 month prior to screening need not be excluded if they satisfy other eligibility criteria.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject or caregiver is an immediate family member or employee of the participating Investigator, any of the participating site staff or GSK staff.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2009-11-02 (Actual); Primary Completion 2010-11-10 (Actual); Study Completion 2010-11-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (Day 1) in the executive function/working memory composite score in the Cog State battery at Week 16 | Baseline (Day 1) and Week 16
  Executive function/working memory composite score was calculated from the three tasks controlled oral word association (a measure of language fluency, planning and working memory where participants were instructed to generate as many as words as they could think of beginning with a specific letter in one minute. They were then requested to do exactly the same for two furthers letters and a score was given for this activity accuracy), category naming (a measure of semantic fluency, planning and working memory where participants were required to generate as many exemplars of the category 'animals' as they could in one minute), and one-back (a valid measure of working memory where participants were shown a single stimulus of a card in the center of the computer screen and were asked for YES" or "NO" to match the current card with the previous card and the accuracy was noted). Change from Baseline is the value at indicated time point minus the Baseline value.
Change from Baseline (Day 1) in the episodic memory composite score in the CogState battery at Week 16 | Baseline (Day 1) and Week 16
  Episodic memory composite score was calculated from the three tasks International Shopping List Task (ISLT) immediate recall, ISLT delayed recall, and Paired Associate Learning (PAL). The Total Score was calculated by taking the mean of all individual task scores. Change from Baseline is the value at indicated time point minus the Baseline value.

SECONDARY OUTCOMES:
Change from Baseline (Day 1) in Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) total score at Weeks 8 and 16 | Baseline (Day 1), Week 8, and 16
  The ADAS-cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place, and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Total scores were calculated as the sum of the individual components. The scale ranges from 0 to 70 with higher scores indicating greater dysfunction. Change from Baseline is the value at indicated time point minus the Baseline value.
Change from Baseline (Day 1) in the attention composite score in the CogState battery at Week 16. | Baseline (Day 1) and Week 16
  Attention composite score was calculated from the two tasks Detection and Identification. If one of the Task Scores used in the calculation of a Composite Score was missing, then the Composite Score was calculated as the mean of the non-missing Task Scores. If more than one Task Score was missing, then the Composite Score was be set to missing. Change from Baseline is the value at indicated time point minus the Baseline value.
Clinician's Interview-Based Impression of Change-plus (CIBIC+) score at Weeks 8 and 16. | At Week 8 and 16
  The term CIBIC+ is also measure of change, though a global assessment of change at screening was collected in addition to the post-randomization visits. However, since the scale is a measure of change itself, change from baseline was not to be calculated. The CIBIC+ global functioning assessment comprises a 7-point rating of severity (assessed at baseline) and change (assessed at subsequent time points). The CIBIC+ assessments were performed by an independent rater. The rater was a trained and experienced neurologist, psychiatrist, neuropsychologist and who does not have access to other participant data for this study. The procedure required separate structured 15-20 minute interviews with the participant and the caregiver.
Change from Baseline (Day 1) to Weeks 8 and 16 of the Disability Assessment for Dementia scale (DAD) total score | Baseline (Day 1), Week 8, and Week 16
  The DAD scale has a total of 40 items. A percentage score was calculated using the formula DAD Percentage Score = 100*(DAD total score / number of item with response). Change from Baseline is the value at indicated time point minus the Baseline value.
Participant's Global Impression of Change (PGIC) score, Carer's Global Impression of Change (CrGIC) score, and Clinician Global Impression of Change (CGIC) at Week 8 and 16 | Week 8 and 16
  Global disease change was also scored by the clinician (CGIC), the caregiver (CrGIC) and the patient (PGIC) using a verbal rating scale. The scale was rated from 1 - 7 (Very much improved, much improved, Minimally improved, No change, minimally worse, much worse, very much worse). No data was available for CGIC parameter at Week 8..
Change from baseline in the Neuropsychiatric Inventory (NPI) at Weeks 8 and 16 | Baseline (Day 1), Week 8, and 16
  NPI is an assessment of the frequency and severity of behavioral disturbances in dementia. The inventory comprises 10 dimensions: delusions, hallucinations, dysphoria, apathy, euphoria, disinhibition, aggressiveness and agitation, irritability, anxiety, and aberrant motor activity. Each dimension has a screening question between 7 and 9 follow-up questions relating to symptoms, asked if the answer to the screening question was 'yes'. The NPI took approximately 10 minutes for the investigator to administer by talking to the caregiver. Change from Baseline is the value at indicated time point minus the Baseline value.
Change from Baseline (Day 1) in Mini Mental State Examination (MMSE) total score at Week 16 | Baseline (Day 1) and Week 16
  The MMSE score scale consists of 11 items covering orientation, memory (recent and immediate), concentration, language and praxis. A Total Score was calculated by adding together the individual items scores. Total Score ranges from 0 to 30, with a lower score indicating greater cognitive impairment. If any item was missing then the total score was set to missing. Change from Baseline is the value at indicated time point minus the Baseline value.
Change from baseline during the titration phase, and to Weeks 8 and 16 of the Pittsburgh Sleep Quality Inventory (PSQI) and Epworth Sleepiness Scale (ESS) | At Week 8 and 16
  The PSQI scale contains 19 self-rated questions from which 7 component scores were calculated; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component was scored on the scale of 0 (no difficulty) to 3 (severe difficulty). The component scores were summed up to produce a Global Score (range 0 to 21). Higher scores indicate worse sleep quality. ESS is an 8-item questionnaire. A total score is calculated by summing the individual item scores. Total scores range from 0 to 24, with higher scores indicating greater sleepiness. Component or item scores were set to missing if any of the individual items used in the calculation of the score were missing. Similarly, the Global Score was set to missing if any of the Component Scores were missing. Change from Baseline was the value at indicated time point minus the Baseline value.
Change from Baseline for Bilateral Score from Olfaction Test at Week 16 | Baseline (Day 1) and Week 16
  The Sniffin' Sticks Screening-12 Test was used for bilateral testing. During the testing, the participant wore a blind fold (a black sleeping mask was supplied with the kit). It was recommended that testing be performed in a well-ventilated room with little or no odor and no disturbances during testing. This test consists of a total of 12 pens and 12 multiple choice answers. Participants were presented with each of the 12 pens at an interval of 30 seconds between each and asked to identify each odorant. For each odorant, the Participant was able to choose from 4 possible answers as to what the smell was. Participants had to identify the item that best described the presented odor. Participants had to choose an item even when they do not perceive an odor or do not feel that their decision was correct. Items identified by participants were noted on the recording sheet. The number of correct answers were recorded. Change from BL is the value at indicated time point minus the BL value
Plasma concentrations of GSK239512 over period | Up to Week 16
  Plasma drug concentration of GSK239512 was analyzed from Week 1 till Week 16 at different doses of 10 mcg, 20 mcg, 40 mcg and 80 mcg. Blood samples for pharmacokinetic analysis of GSK239512 were collected at each clinic visit. Two PK samples were collected; one sample with 15 minutes prior to the start of the CogState Neuropsychological Test Battery (NTB) and one sample within 15 minutes of completion of the CogState NTB.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to 18 weeks
  Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Number of participants with vital signs outside clinical concern range (Systolic blood pressure [SBP], diastolic blood pressure [DBP], and heart rate [HR]) | Up to Week 18
  The SBP was considered as of clinical concern if <90 or >140 millimeters of mercury (mm of Hg) and increase from Baseline more than or equal to (>=) 40 mm Hg occurred. For DBP, Increase from baseline >=30 mm of Hg was considered as of clinical concern. For HR, if the values are <50 beats per minute (bpm) or >100 bpm, and increase from baseline >=30 bpm, it was considered as of clinical concern. All readings were taken in sitting position. The Data has been presented only for abnormal vital signs.
Number of participants with hematological and clinical chemistry parameters outside the reference range up to 16 weeks | Up to 16 weeks
  The data for number of participants with abnormal values; high (H) or low (L) was reported for on-treatment time span. Only the data outside the reference range has been presented. Baseline was considered to be the last available assessment prior to the study drug.
Number of participants with abnormal electrocardiogram (ECG) over period | Up to 18 weeks
  This analysis was accounted for the maximum post-baseline on-treatment QTc observed. Participant was counted once in the most extreme clinical interpretation category they had within a visit. For interpretations, the least to most extreme interpretations were normal; abnormal - not clinically significant; abnormal - clinically significant. The Baseline value was based on the mean of the screening assessment values. ECG measurements were collected on paper or electronically at each investigational center. Only the abnormal values were presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- Bulgaria (2):
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- Chile (3):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Czechia (3):
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Trutnov
- Germany (7):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
- Russia (7):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Slovakia (3):
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Levoča
  - GSK Investigational Site, Michalovce
- South Korea (2):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- United Kingdom (3):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110651 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register